CLINICAL TRIAL: NCT03331835
Title: A Phase 4 Trial Comparing the Efficacy of Subcutaneous Injections of Brodalumab to Oral Administrations of Fumaric Acid Esters in Adults With Moderate to Severe Plaque Psoriasis
Brief Title: A Trial Comparing the Efficacy of Subcutaneous Injections of Brodalumab to Oral Administrations of Fumaric Acid Esters in Adults With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0160-1327; 2016-003867-21 (EudraCT Number)
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2020-02

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — brodalumab; Fumarates; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brodalumab (Experimental): Kyntheum® (brodalumab)
  pre-filled syringe 210 mg/1.5 mL solution for subcutaneous injections.
  First 3 injections are administered weekly, and hereafter every two weeks (Q2W).
  Interventions: Biological: Brodalumab
- Fumaric acid esters (Active Comparator): Fumaderm® initial dose tablets (30 mg dimethyl fumarate, 67 mg ethyl hydrogen fumarate calcium salt, 5 mg ethyl hydrogen fumarate magnesium salt, 3 mg ethyl hydrogen fumarate zinc salt)
  Fumaderm® tablets (120 mg dimethyl fumarate, 87 mg ethyl hydrogen fumarate calcium salt, 5 mg ethyl hydrogen fumarate magnesium salt, 3 mg ethyl hydrogen fumarate zinc salt)
  Fumaderm® tablets are administered orally up to 3 times daily in accordance with the dosing scheme in the label.
  Interventions: Drug: Fumaric acid esters

INTERVENTIONS:
Biological: Brodalumab — Brodalumab is a recombinant fully human monoclonal immunoglobulin IgG2-antibody that binds with high affinity to human interleukin 17 receptor A (IL-17RA).
  Blocking IL-17RA inhibits IL-17 cytokine-induced responses and results in reduced or normalised inflammation of the skin in subjects with psoriasis.
  Other Names: Kyntheum®
  Arms: Brodalumab
Drug: Fumaric acid esters — Fumaric acid esters have been used to treat psoriasis since 1959. Systemic therapy with fumaric acid esters is based on an established dosing scheme with a gradual increase to improve tolerability, especially with regards to gastrointestinal side effects.
  Other Names: Fumaderm®
  Arms: Fumaric acid esters

SUMMARY:
The primary objective is to demonstrate added benefit of brodalumab versus a selected systemic comparator in treatment of moderate to severe plaque psoriasis in Germany in subjects who have not previously received systemic treatment for psoriasis.

Fumaric acid esters have been selected as the comparator because it is an established systemic treatment of psoriasis in Germany.

DETAILED DESCRIPTION:
A 24-week, randomised, open-label, active-controlled, parallel group, multi-centre trial with investigator-blinded efficacy assessments

ELIGIBILITY:
Main Criteria for Inclusion:

* Men or women ≥18 years of age at the time of screening.
* Subjects with chronic plaque type psoriasis diagnosed at least 6 months before randomisation.
* Subjects with moderate to severe plaque psoriasis in whom topical therapy is not adequate and who are candidates for systemic therapy, defined at randomisation by PASI 10, affected BSA >10%, and DLQI >10.
* Subject has no known history of active tuberculosis.
* Subject has a negative test for tuberculosis taken at screening (negative Quantiferon test).
* Subject and/or subject's designee is/are capable of administering subcutaneous injections.

Main Criteria for Exclusion:

* Previous or current systemic treatment of plaque psoriasis or known contraindication for systemic therapy.
* Previous or current PUVA (psoralens and ultraviolet A) therapy.
* Washouts and non-permitted drugs:

  1. Have received phototherapy (UVA light therapy without psoralens, UVB light therapy, excimer laser, tanning beds etc. within 4 weeks of baseline, or
  2. Have had topical psoriasis treatment within 2 weeks of baseline (exceptions: bland emollients without urea or beta or alpha hydroxy acids)
  3. Have received any biologic immune modulating treatments used for indication other than psoriasis within 4 weeks of baseline or within a period of 5 half-lives of the IMP, whichever is longer
  4. Have received any other systemic immune modulating treatment (including but not limited to oral retinoids, methotrexate, calcineurin inhibitors, oral or parenteral corticosteroids etc. used for indications other than psoriasis) within 4 weeks of baseline or within a period of 5 half-lives of the IMP, whichever is longer.
* Subjects with any of the following laboratory abnormalities at screening:

  1. Leukocyte cell count below 3×10^9/L or lymphocyte count below 0.7×10^9/L
  2. Aspartate aminotransferase (AST) or alanine transferase (ALT) > 2× ULN (upper level of normal limit)
  3. Absolute neutrophil count < 2×10^9/L
  4. Serum creatinine > ULN.
* History of depressive disorder within the last 2 years including current antidepressive treatment.
* Subjects with a history of suicidal behaviour (suicide attempt).
* Any suicidal ideation of severity 4 or 5 based on the eC-SSRS questionnaire at screening.
* A PHQ-8 score of ≥10 corresponding to moderate to severe depression at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (30):
- Germany (30):
  - Fachklinik Bad Bentheim Klinik für Dermatologie, Bad Bentheim
  - Charité - Universitätsmedizin Berlin Klinik für Dermatologie, Venerologie und Allergologie Psoriasis Studien Zentrum, Berlin
  - Rothhaar Studien GmbH Dermatologisches Studienzentrum, Berlin
  - Hautarztpraxis Dr. Wildfeuer, Berlin
  - Klinikum Bielefeld Klinik für Dermatologie und Allergologie, Bielefeld
  - Hauttumorzentrum Ruhr- Universität im St. Josef Hospital, Bochum
  - Hautarztpraxis Dr. Niesmann und Dr. Othlinghaus, Bochum
  - Universitätsklinikum Bonn (AöR) Klinik und Poliklinik für Dermatologie und Allergologie, Bonn
  - Elbe Klinikum Buxtehude Klinik für Dermatologie, Buxtehude
  - Rosenpark Research, Darmstadt
  - Universitätsklinikum Carl Gustav Carus Klinik und Poliklinik für Dermatologie, Dresden
  - Universitätsklinikum Erlangen Hautklinik, Erlangen
  - Universitätsklinikum Frankfurt Klinik für Dermatologie, Frankfurt
  - Derma-Study-Center-Friedrichshafen, Friedrichshafen
  - Gemeinschaftspraxis Rotterdam & Kollegen Facharzt für Haut & Geschlechtskrankheiten, Gelsenkirchen
  - Universitätsklinikum Hamburg-Eppendorf, Institut für Versorgungsforschung in der Dermatologie und bei Pflegeberufen, Hamburg
  - SCIderm GmbH, Hamburg
  - Medizinische Hochschule Hannover Klinik für Dermatologie Allergologie und Venerologie, Hanover
  - Universitäts-Hautklinik Heidelberg, Heidelberg
  - Klinik für Dermatologie, Venerologie und Allergologie Universitätsklinikum Schleswig-Holstein, Campus Kiel Psoriasis-Zentrum, Kiel
  - Exellenzzentrum Entzündungsmedizin (CCIM) Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - University Medical Center Mainz Department of Dermatology and Allergy, Clinical Research Center, Mainz
  - Universitätsklinikum Mannheim der Universität Heidelberg Klinik für Dermatologie, Venerologie und Allergologie, Mannheim
  - Technische Universität München Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Klinische Forschung Osnabrück - Klifos, Osnabrück
  - KLINIKUM VEST GmbH Knappschaftskrankenhaus Recklinghausen Klinik für Dermatologie und Allergologie, Recklinghausen
  - Gemeinschaftspraxis Weber & Crainic, Schweinfurt
  - Hautarztpraxis Dres. Leitz, Stuttgart
  - University Medical Center University of Tübingen, Tübingen
  - Hautarztpraxis, Witten

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fumaric Acid Esters: Fumaderm® initial dose tablets (30 mg dimethyl fumarate, 67 mg ethyl hydrogen fumarate calcium salt, 5 mg ethyl hydrogen fumarate magnesium salt, 3 mg ethyl hydrogen fumarate zinc salt). Fumaderm® tablets (120 mg dimethyl fumarate, 87 mg ethyl hydrogen fumarate calcium salt, 5 mg ethyl hydrogen fumarate magnesium salt, 3 mg ethyl hydrogen fumarate zinc salt).
  Fumaderm® tablets are administered orally up to 3 times daily in accordance with the dosing scheme in the label.
Period: Overall Study
Arm/Group | Brodalumab | Fumaric Acid Esters
Started | 105 | 105
Completed | 91 | 58
Not Completed | 14 | 47

BASELINE CHARACTERISTICS:
Groups:
- Brodalumab: Subcutaneous (s.c.) brodalumab 210 mg once weekly at Weeks 0, 1, and 2, and 210 mg s.c. every 2 weeks.
- Fumaric Acid Esters: Oral fumaric acid esters up to 240 mg 3 times daily (TID).
- Total: Total of all reporting groups
Arm/Group | Brodalumab | Fumaric Acid Esters | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 97 | 193
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 73 | 72 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 100 | 103 | 203
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 104 | 105 | 209
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 105 | 105 | 210
Height [Mean (Standard Deviation); unit: cm] | 175 (9.6) | 176 (9.8) | 175 (9.7)
Weight [Mean (Standard Deviation); unit: kg] | 87.8 (20.4) | 86.6 (21.1) | 87.2 (20.7)
Mean weight in participants weighing <100 kg [Mean (Standard Deviation); unit: kg] — Population: Not all participants weighed below 100 kg. This section shows the mean weight of participants weighing less than 100 kg.
  kg
    number analyzed (Participants) | 79 | 79 | 158
    (all) | 78.4 (11.9) | 77.2 (12.8) | 77.8 (12.4)
Mean weight in participants weighing >=100 kg [Mean (Standard Deviation); unit: kg] — Population: Not all participants weighed over 100 kg. This section shows the mean weight of participants equal to or more than 100 kg
  kg
    number analyzed (Participants) | 26 | 26 | 52
    (all) | 116 (13.2) | 115 (13.9) | 116 (13.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (5.7) | 28.0 (6.0) | 28.2 (5.9)
Duration of psoriasis [Mean (Standard Deviation); unit: years] | 14.3 (11.5) | 13.2 (11.7) | 13.7 (11.6)
PASI score [Mean (Standard Deviation); unit: score on a scale] — The psoriasis area and severity index (PASI) score grades the extent and severity of psoriatic involvement for each of four body regions (head and neck, upper extremities, trunk, and lower extremities) using a 7-point scale for extent of involvement in each body region and 5-point scales for severity of each of the clinical signs redness, thickness, and scaliness in each body region.
  Psoriasis Area and Severity Index is a scale ranging from 0 (no disease) to 72 (maximal disease).
  score on a scale | 17.2 (5.9) | 17.8 (6.7) | 17.5 (6.3)
sPGA score [Mean (Standard Deviation); unit: score on a scale] — The static Physicians Global Assessment (sPGA) is a 6-point scale that represents the average lesion severity on the trunk and limbs. The assessment is based on the condition of the disease at the time of evaluation.
  Static Physician's Global Assessment is a scale ranging rom 0 (clear skin) to 5 (severe disease).
  score on a scale | 3.5 (0.6) | 3.5 (0.7) | 3.5 (0.6)
BSA score [Mean (Standard Deviation); unit: score on a scale] | 24.8 (15.2) | 25.5 (14.9) | 25.2 (15.1)
NAPSI score [Mean (Standard Deviation); unit: score on a scale] — The Nail Psoriasis Severity Index (NAPSI) grades nails by dividing the nail area into 4 quarters. The following 8 clinical features of nail psoriasis are then scored based on the number of quarters in which the feature is present (0 to 4) to arrive at a NAPSI score of 0 to 32 for each nail:
  * Pitting.
  * Leukonychia.
  * Red spots in lunula.
  * Nail plate crumbling.
  * Oil drop (salmon patch) discoloration.
  * Onycholysis.
  * Nail bed hyperkeratosis.
  * Splinter haemorrhages.
  A negative change in NAPSI score means that the NAPSI score was lower at the time of data collection. Population: Not all participants had nail involvement at baseline. Only participants with nail involvement at baseline were included here.
  score on a scale
    number analyzed (Participants) | 43 | 38 | 81
    (all) | 6.4 (4.4) | 7.7 (4.9) | 7.0 (4.7)
DLQI score [Mean (Standard Deviation); unit: score on a scale] — The Dermatology Life Quality Index (DLQI) consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4 point Likert scale (0 = not at all ⁄not relevant; 1 = a little; 2 = a lot; 3 = very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor QoL.
  score on a scale | 18.8 (5.2) | 18.5 (4.9) | 18.7 (5.1)
PSI score [Mean (Standard Deviation); unit: score on a scale] — The Psoriasis Symptom Inventory (PSI) consists of eight psoriasis-specific questions. Trial participants rated the severity of their symptoms in the last 24 hours from 'not at all' to 'very severe,' ranging from 0 to 4. Total scores range from 0 to 32 with higher scores indicating worse symptoms. PSI response is defined as total score ≤8 and no item score >1. Symptom-free day is defined as having daily total PSI of 0 on that day. Population: Not all subjects had a baseline PSI measurement.
  score on a scale
    number analyzed (Participants) | 83 | 78 | 161
    (all) | 14.8 (5.4) | 17.9 (5.3) | 16.3 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Having Least 75% Lower Psoriasis Area and Severity Index (PASI) Score Relative to Baseline (PASI 75 Response) From Baseline at Week 24
Description: The PASI score grades the extent and severity of psoriatic involvement for each of four body regions (head and neck, upper extremities, trunk, and lower extremities) using a 7-point scale for extent of involvement in each body region and 5-point scales for severity of each of the clinical signs redness, thickness, and scalliness in each body region.
  Psoriasis Area and Severity Index is a scale ranging from 0 (no disease) to 72 (maximal disease).
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 105 | 105
Participants | 85 | 40
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; Estimated risk difference, 95% CI and p-value are derived from Cochran-Mantel-Haenszel (CMH) analysis stratified by weight group at baseline (≤100 kg, > 100 kg). Non-responder Imputation (NRI) was used to impute missing data. Treatment groups were defined as randomised treatment; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 95% CI and p-value are derived from CMH analysis stratified by weight group at baseline (≤100 kg, > 100 kg); Risk Difference (RD) = 42.86, 95% CI 2-sided [30.93 to 54.79]

2. Primary Outcome: Static Physician's Global Assessment (sPGA) Scale Score of 0 or 1 at Week 24
Description: sPGA is a 6-point scale that represents the average lesion severity on the trunk and limbs. The assessment is based on the condition of the disease at the time of evaluation.
  Static Physician's Global Assessment is a scale ranging rom 0 (clear skin) to 5 (severe disease).
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 105 | 105
Participants | 68 | 21
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 95% CI and p-value are derived from CMH analysis stratified by weight group at baseline (≤100 kg, > 100 kg); Risk Difference (RD) = 44.76, 95% CI 2-sided [32.81 to 56.71]

3. Secondary Outcome: Having Least 90% Lower Psoriasis Area and Severity Index (PASI) Score Relative to Baseline (PASI 90 Response) From Baseline at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 105 | 105
Participants | 69 | 23
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 43.81, 95% CI 2-sided [31.78 to 55.84]

4. Secondary Outcome: Having 100% Lower Psoriasis Area and Severity Index (PASI) Score Relative to Baseline (PASI 100 Response) From Baseline at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 105 | 105
Participants | 42 | 9
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 31.43, 95% CI 2-sided [20.76 to 42.10]

5. Secondary Outcome: Change From Baseline at Week 24 in PASI Score
Description: The PASI score grades the extent and severity of psoriatic involvement for each of four body regions (head and neck, upper extremities, trunk, and lower extremities) using a 7-point scale for extent of involvement in each body region and 5-point scales for severity of each of the clinical signs redness, thickness, and scalliness in each body region. Psoriasis Area and Severity Index is a scale ranging from 0 (no disease) to 72 (maximal disease).
  A negative change in PASI score means that the PASI score was lower at the time of data collection.
Time Frame: Baseline to Week 24
Population: The number of analysed participants is not the same as the number of randomised participants, as participants with missing data in all visits for a given endpoint are not included in the mixed model for repeated measurements (MMRM) analysis used to analyse the endpoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 100 | 96
score on a scale | -15.69 (0.59) | -12.62 (0.67)
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; The endpoint was analysed using mixed model for repeated measures (MMRM) model including treatment group, week, interaction between treatment and time, baseline value, and baseline weight group as fixed factors. Within participant covariance was estimated by an unstructured covariance matrix. Treatment groups were defined as randomised treatment; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -3.08, 95% CI 2-sided [-4.83 to -1.33]

6. Secondary Outcome: Percent Change From Baseline in PASI Score at Week 24
Description: The PASI score grades the extent and severity of psoriatic involvement for each of four body regions (head and neck, upper extremities, trunk, and lower extremities) using a 7-point scale for extent of involvement in each body region and 5-point scales for severity of each of the clinical signs redness, thickness, and scalliness in each body region. Psoriasis Area and Severity Index is a scale ranging from 0 (no disease) to 72 (maximal disease).
  A negative value in the percent change from baseline that the PASI score was lower at the time of data collection.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percent change in PASI
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 100 | 96
percent change in PASI | -90.03 (2.25) | -73.67 (2.63)
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -16.36, 95% CI 2-sided [-23.03 to -9.68]

7. Secondary Outcome: Change From Baseline at Week 24 in Affected Body Surface Area (BSA)
Description: The surface area of the participant's hand (palm and fingers) is used as a reference measurement to calculate the percentage of each body region that is affected by psoriasis. One hand is approximately equal to 1% total BSA.
  Furthermore, the complete body surface area (BSA=100%) can be divided into regions that approximates percentages of BSA as follows: head and neck (10%), upper extremities (20%), the trunk including the axillae and groin (30%), and finally the lower extremities, including the buttocks (40%).
  A negative value in the percent change from baseline that the affected BSA was lower at the time of data collection.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 105 | 105
percent change | -20.82 (1.48) | -11.91 (1.48)
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -8.91, 95% CI 2-sided [-13.00 to -4.81]

8. Secondary Outcome: Psoriasis Symptom Inventory (PSI) Responder at Week 24 (Total Score ≤ 8, With no Item Scores > 1)
Description: The PSI consists of eight psoriasis-specific questions. Trial participants rated the severity of their symptoms in the last 24 hours from 'not at all' to 'very severe,' ranging from 0 to 4. Total scores range from 0 to 32 with higher scores indicating worse symptoms. PSI response is defined as total score ≤8 and no item score >1. Symptom-free day is defined as having daily total PSI of 0 on that day.
Time Frame: Week 24
Population: PSI data was missing for many participants at baseline and Week 24. For this reason, no statistical analysis was performed. The data shown is therefore descriptive data.
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 23 | 15
Participants | 15 | 13

9. Secondary Outcome: PSI Total Score of 0 at Week 24
Description: as for outcome 8
Time Frame: Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 23 | 15
Participants | 5 | 3

10. Secondary Outcome: Number of Symptom-free Days From Randomisation to Week 24
Description: as for outcome 8
Time Frame: Baseline to Week 24
Population: PSI data was missing for many participants at baseline and Week 24. For this reason, no statistical analysis was performed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 64 | 33
days | 0.44 (0.8) | 0.42 (1.3)

11. Secondary Outcome: Burden of Symptoms
Description: Burden of symptoms was assessed as the normalised area under the curve (AUC) of PSI from baseline to the last available assessment. The AUC for the PSI total score was calculated for each participant using the standard trapezoidal rule. The AUC was normalised by dividing it with the time from baseline to the last available assessment of the PSI total score.
  The PSI consists of eight psoriasis-specific questions. Trial participants rated the severity of their symptoms in the last 24 hours from 'not at all' to 'very severe,' ranging from 0 to 4. Total scores range from 0 to 32 with higher scores indicating worse symptoms.
Time Frame: Baseline to Week 24
Population: Not all participants had recorded PSI data, therefore the analysed number of participants is lower than the randomised number of participants.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 83 | 78
score on a scale | 6.00 (0.54) | 10.92 (0.55)
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; The AUC was analysed using analysis of covariance (ANCOVA) with treatment group, baseline weight group, and the baseline PSI total score as explanatory variables. Treatment groups are defined as randomised treatment; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -4.92, 95% CI 2-sided [-6.31 to -3.53]

12. Secondary Outcome: Change From Baseline at Week 24 in Dermatology Life Quality Index (DLQI) Total Score
Description: DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4 point Likert scale (0 = not at all ⁄not relevant; 1 = a little; 2 = a lot; 3 = very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor QoL.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 99 | 86
score on a scale | -16.67 (0.61) | -14.10 (0.70)
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; The endpoint is analysed by using mixed model for repeated measurements (MMRM) model including treatment group, week, interaction between treatment and time, baseline value, and baseline weight group as fixed factors. Within participant covariance was estimated by an unstructured covariance matrix. Treatment groups are defined as randomised treatment; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Net) = -2.57, 95% CI 2-sided [-4.32 to -0.82]

13. Secondary Outcome: DLQI Total Score of 0 or 1 at Week 24
Description: DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their QoL over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4 point Likert scale (0 = not at all ⁄not relevant; 1 = a little; 2 = a lot; 3 = very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor QoL.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 105 | 105
Participants | 70 | 27
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; Test type: Superiority — Estimated risk difference, 95% CI and p-value are derived from Cochran-Mantel-Haenszel (CMH) analysis stratified by weight group at baseline (<=100 kg, > 100 kg). Non-responder Imputation (NRI) was used to impute missing data. Treatment groups were defined as randomised treatment; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 40.95, 95% CI 2-sided [28.75 to 53.16]

14. Other Pre Specified Outcome: Change From Baseline at Week 24 in NAPSI Total Score
Description: The Nail Psoriasis Severity Index (NAPSI) grades nails by first dividing the nail area with imaginary horizontal and vertical lines into 4 quarters. The following 8 clinical features of nail psoriasis are then scored based on the number of quarters in which the feature is present (0 to 4) to arrive at a NAPSI score of 0 to 32 for each nail:
  * Pitting.
  * Leukonychia.
  * Red spots in lunula.
  * Nail plate crumbling.
  * Oil drop (salmon patch) discoloration.
  * Onycholysis.
  * Nail bed hyperkeratosis.
  * Splinter haemorrhages.
  A negative change in NAPSI score means that the NAPSI score was lower at the time of data collection.
Time Frame: Baseline to Week 24
Population: Only participants with nail involvement at baseline were included in the analysis. Therefore the number of analysed participants differs from the number of randomised participants.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Brodalumab | Fumaric Acid Esters
Number analyzed (Participants) | 43 | 38
score on a scale | -2.97 (0.54) | -1.26 (0.57)
Statistical Analysis 1: Comparison: Brodalumab vs Fumaric Acid Esters; Test type: Superiority — The endpoint was analysed by using mixed model for repeated measures (MMRM) model including treatment group, week, interaction between treatment and time, baseline value, and baseline weight group as fixed factors. Within participant covariance was estimated by an unstructured covariance matrix. Treatment groups were defined as randomised treatment; p = 0.028, Mixed Models Analysis; Mean Difference (Net) = -1.72, 95% CI 2-sided [-3.24 to -0.19]

ADVERSE EVENTS:
Time Frame: From the first day of investigational medicinal product (IMP) administration and until 32 weeks later for brodalumab and 26 weeks later for fumaric acid esters. The difference in collection periods was due to the different half-lives of the IMPs.
Groups:
- Brodalumab 210 mg: Kyntheum® (brodalumab) pre-filled syringe 210 mg/1.5 mL solution for subcutaneous injections. First 3 injections are administered weekly, and hereafter every two weeks (Q2W).
- Fumaric Acid Ester: Fumaderm® initial dose tablets (30 mg dimethyl fumarate, 67 mg ethyl hydrogen fumarate calcium salt, 5 mg ethyl hydrogen fumarate magnesium salt, 3 mg ethyl hydrogen fumarate zinc salt) > Fumaderm® tablets (120 mg dimethyl fumarate, 87 mg ethyl hydrogen fumarate calcium salt, 5 mg ethyl hydrogen fumarate magnesium salt, 3 mg ethyl hydrogen fumarate zinc salt).
  Fumaderm® tablets are administered orally up to 3 times daily in accordance with the dosing scheme in the label.
Arm/Group | Brodalumab 210 mg | Fumaric Acid Ester
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/102
Serious Adverse Events (participants affected / at risk) | 3/104 | 1/102
Other Adverse Events (participants affected / at risk) | 66/104 | 90/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brodalumab 210 mg (N=104) | Fumaric Acid Ester (N=102)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reactive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brodalumab 210 mg (N=104) | Fumaric Acid Ester (N=102)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 11 (13)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 28 (43)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 59 (77)
Nausea (Gastrointestinal disorders) | 6 (7) | 9 (13)
Fatigue (General disorders) | 5 (6) | 6 (8)
Viral upper respiratory tract infection (Infections and infestations) | 35 (41) | 21 (24)
Overdose (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Headache (Nervous system disorders) | 13 (27) | 12 (19)
Depressive symptom (Psychiatric disorders) | 5 (5) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 29 (40)

LIMITATIONS AND CAVEATS:
Operational challenges with the ePRO diary device given to trial participants led to missing data at baseline and Week 24. This made the analyses of the secondary patient-reported endpoints PSI response rate and PSI total score of 0 or 1 impossible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators have agreed to refrain from publishing based on data from this trial until the multi-center publication containing data from all sites has been published (usually after approx. 18 months). After this, any publication by individual investigators must be reviewed by the sponsor prior to submission. Sponsor has the right to remove any commercially confidential information and/or delay the publication up to 4 months to allow time for activities protecting intellectual rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT03331835/Prot_SAP_000.pdf